CLINICAL TRIAL: NCT05898815
Title: A Multicenter Study of Retrospective Rehabilitation Medical Data for the Development for Medical Twins
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bundang CHA Hospital (Other)
Responsible Party: Principal Investigator, MinYoung Kim, MD, PhD, Bundang CHA Hospital, Bundang CHA Hospital
Other Study IDs: 2021-11-020
Record Dates: First submitted 2023-05-23; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Health-Related Behavior; Stroke
MeSH Terms: conditions — Health Behavior; Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy subjects and stroke patients: Healthy subjects and stroke patients
  Interventions: Diagnostic Test: Medical record collection

INTERVENTIONS:
Diagnostic Test: Medical record collection — Medical record collection

SUMMARY:
Based on previous studies, when medical digital twin-based convergence medical contents are applied to degenerative musculoskeletal and central nervous system diseases, it is possible to more accurately evaluate the subject's motor function and neurological function to predict the subject's disease. In order to create an effective ICT application protocol and clinically apply a treatment program that can improve the subject's kinematic function and neurological function, etc.

ELIGIBILITY:
1. Inclusion Criteria:

   * Healthy subjects : who underwent imaging examination at Bundang CHA hospital from January 1, 2010 to December 31, 2021
   * Stroke patients : who underwent imaging examination at Bundang CHA hospital from January 1, 2010 to December 31, 2021
2. Exclusion criteria - Who cannot meet the inclusion criteria

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy and stroke patients
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-12-22 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Imaging examination | A time point at which imaging was performed between January 1, 2010 and December 31, 2021
  The results of X-ray measurement in whole spin AP and lateral, low extremty AP & lateral, foot AP & lateral, The results of multispine computed tomography of C-spine, T-spin and L-spine without CM, The results of magnetic resonance imaging of brain MRI and diffusion tensor imaging tractography

SECONDARY OUTCOMES:
Basic characteristics | A time point at which imaging was performed between January 1, 2010 and December 31, 2021
  Sex, age, stroke onset, stroke diagnosis, history

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Rehabilitation Medicine, CHA Bundang Medical Center, Seongnam, South Korea

IPD SHARING:
Plan to Share IPD: Yes